CLINICAL TRIAL: NCT01772290
Title: A Clinical Drug-Drug Interaction Study to Evaluate the Effect of a Proton Pump Inhibitor, a Combined P-gp/CYP3A4 Inhibitor, and a CYP2C9 Inhibitor on the Pharmacokinetics of Vismodegib
Brief Title: A Drug-Drug Interaction Study of the Effect of Rabeprazole, Itraconazole or Fluconazole on the Pharmacokinetics of Vismodegib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GP28465
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Fluconazole; Itraconazole; Rabeprazole; HhAntag691

ARMS (4):
- A: Vismodegib (Active Comparator)
  Interventions: Drug: vismodegib
- B: Rabeprazole + Vismodegib (Experimental)
  Interventions: Drug: rabeprazole; Drug: vismodegib
- C: Itraconazole + Vismodegib (Experimental)
  Interventions: Drug: itraconazole; Drug: vismodegib
- D: Fluconazole + Vismodegib (Experimental)
  Interventions: Drug: fluconazole; Drug: vismodegib

INTERVENTIONS:
Drug: fluconazole — Multiple oral doses
  Arms: D: Fluconazole + Vismodegib
Drug: itraconazole — Multiple oral doses
  Arms: C: Itraconazole + Vismodegib
Drug: rabeprazole — Multiple oral doses
  Arms: B: Rabeprazole + Vismodegib
Drug: vismodegib — Multiple oral doses

SUMMARY:
This randomized, open-label, 4-arm, multiple-dose study will evaluate the effect of coadministration of a protein pump inhibitor, an inhibitor of P-glycoprotein and CYP3A4, or an inhibitor of CYP2C9 on the pharmacokinetics of vismodegib in healthy female subjects of non-childbearing potential. Subjects will be randomized to receive multiple oral doses of vismodegib, alone or in combination with multiple oral doses of either rabeprazole, itraconazole or fluconazole. Anticipated time on study treatment is up to 11 days.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential
* Body mass index (BMI) 18 to 32 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, physical examination. 12-lead ECG, and vital signs
* Clinical laboratory evaluations, complete blood count and urinalysis within the normal range for the test laboratory, unless not deemed clinically significant by the investigator
* Negative test for drugs of abuse at screening and check-in (including alcohol)
* Negative for hepatitis B, hepatitis C and HIV infection
* Non-childbearing potential is defined as: non-pregnant, non-lactating, and either postmenopausal for at least 1 year or surgically sterile (e.g. bilateral oophorectomy and/or hysterectomy)

Exclusion Criteria:

* Significant history or clinical evidence of any metabolic (including type 1 or 2 diabetes). allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, endocrine, GI (including gastric or duodenal ulcers), Zollinger-Ellison syndrome, Barrett's esophagus, urological, neurological, or psychiatric disorder
* History of inflammatory arthritis
* History of symptomatic hypotension
* History of seizure disorders
* History of bipolar or major depressive disorder
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (appendectomy, hernia repair, and/or cholecystectomy will be allowed)
* History of alcoholism or drug addiction within 1 year prior to check-in
* Use of any tobacco- or nicotine-containing products within 6 months prior to check-in
* Participation in any other investigational study drug or biological agent trial in which receipt of investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to check-in
* Use of PPIs, H2-receptor antagonists, or antacids within 1 month prior to check-in
* History of chronic PPI use (> 30 days of continuous daily dosing) within 6 months of check-in

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Relative effect of rabeprazole on steady-state pharmacokinetics of vismodegib: Area under the concentration-time curve (AUC)/Steady-state concentration (Css) | up to 12 days
Relative effect of itraconazole on steady-state pharmacokinetics of vismodegib: Area under the concentration-time curve (AUC)/Steady-state concentration (Css) | up to 12 days
Relative effect of fluconazole on the steady-state pharmacokinetics of vismodegib: Area under the concentration-time curve (AUC)/Steady-state concentration (Css) | up to 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (2):
- United States (2):
  - Daytona Beach, Florida
  - Dallas, Texas

REFERENCES:
- [Derived] Malhi V, Colburn D, Williams SJ, Hop CE, Dresser MJ, Chandra P, Graham RA. A clinical drug-drug interaction study to evaluate the effect of a proton-pump inhibitor, a combined P-glycoprotein/cytochrome 450 enzyme (CYP)3A4 inhibitor, and a CYP2C9 inhibitor on the pharmacokinetics of vismodegib. Cancer Chemother Pharmacol. 2016 Jul;78(1):41-9. doi: 10.1007/s00280-016-3020-z. Epub 2016 May 6. PMID 27154174